CLINICAL TRIAL: NCT00256932
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase 3 Study to Evaluate the Efficacy and Safety of Alvimopan 0.5mg Once Daily and 0.5mg Twice Daily for 12 Weeks for the Treatment of Opioid-Induced Bowel Dysfunction in Adults Taking Opioid Therapy for Persistent Non-Cancer Pain
Brief Title: Treatment Of Constipation Due To Opioids Being Taken For Persistent Non-Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-767905/012
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2011-12

CONDITIONS: Bowel Dysfunction; Constipation
Keywords: bowel dysfunction; constipation; gastrointestinal; opioids; pain; non-cancer pain; Opioid-induced
MeSH Terms: conditions — Intestinal Diseases; Constipation; Pain | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Alvimopan 0.5 mg once daily (Experimental)
  Interventions: Drug: alvimopan
- alvimopan 0.5 mg twice daily (Experimental)
  Interventions: Drug: alvimopan

INTERVENTIONS:
Drug: alvimopan — 0.5 mg
  Other Names: Entereg
  Arms: Alvimopan 0.5 mg once daily; alvimopan 0.5 mg twice daily
Drug: Placebo
  Arms: Placebo

SUMMARY:
Adults who are taking opioid therapy for persistent non-cancer pain and have resulting opioid-induced bowel dysfunction (OBD) will be randomized (1:1:1) to one 2 alvimopan arms, or to placebo. The primary objective of this phase 3 confirmatory study is to compare alvimopan with placebo for efficacy in the treatment of OBD. The primary efficacy endpoint is based on frequency of bowel movements. Subjects will be required to: (1) track their bowel movements and other bowel symptoms and (2) attend 6 clinic visits over 4 months.

ELIGIBILITY:
Inclusion criteria:

* Has consented to participate in this study.
* Taking opioid therapy for persistent non-cancer pain.
* Has bowel dysfunction mainly due to opioids.
* Has bowel dysfunction since starting opioids as defined by infrequent bowel movements and additional bowel-related symptoms.
* Willing to discontinue laxative therapy (will be provided study-specific standardized laxative if needed).
* Willing to report daily bowel symptoms.

Exclusion criteria:

* Pregnant, lactating, or planning to become pregnant.
* Not ambulatory.
* Participated in another trial with an investigational drug in the past 30 days.
* Taking opioids for the management of drug addiction or cancer-related pain.
* Severe constipation whereby the subject is at immediate risk of developing serious complications of constipation.
* Gastrointestinal or pelvic disorders known to affect bowel transit, produce gastrointestinal (GI) obstruction, or contribute to bowel dysfunction.
* HIV-infected, has active hepatitis, or has ever been infected with hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2005-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
to compare alvimopan with placebo for efficacy in the treatment of OBD

SECONDARY OUTCOMES:
Safety and tolerability, quality of life, pharmacokinetics, pharmacogenetics (dependent on results from other data)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (171):
- United States (117):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Calera, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Tallassee, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Beuna Park, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Brooksville, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Meyers, Florida
  - GSK Investigational Site, Gainsville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Niceville, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Dawsonville, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Bloomington, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Fenton, Missouri
  - GSK Investigational Site, Manchester, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Incline Village, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valley Stream, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Concord, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Nazareth, Pennsylvania
  - GSK Investigational Site, Whitehall, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Woonsocket, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Brownwood, Texas
  - GSK Investigational Site, Colleyville, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Lacey, Washington
  - GSK Investigational Site, Spokane, Washington
- GSK Investigational Site, Vienna, Austria
- Canada (12):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Denmark (3):
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Ishøj
  - GSK Investigational Site, Odense C
- GSK Investigational Site, Tallinn, Estonia
- GSK Investigational Site, Helsinki, Finland
- Germany (19):
  - GSK Investigational Site, Fellbach, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Pinneberg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Cork, Ireland
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Wroclaw
- United Kingdom (13):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Slough, Berkshire
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Ashford, Middlesex
  - GSK Investigational Site, Sunbury-on-Thames, Middlesex
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Bexhill-on-Sea, East Sussex
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Yaxley, Peterborough
  - GSK Investigational Site, York

REFERENCES:
- [Result] Jansen JP, Lorch D, Langan J, Lasko B, Hermanns K, Kleoudis CS, Snidow JW, Pierce A, Wurzelmann J, Mortensen ER. A randomized, placebo-controlled phase 3 trial (Study SB-767905/012) of alvimopan for opioid-induced bowel dysfunction in patients with non-cancer pain. J Pain. 2011 Feb;12(2):185-93. doi: 10.1016/j.jpain.2010.06.012. PMID 21292169